CLINICAL TRIAL: NCT03438851
Title: Assessing Neurophysiological Changes in Individuals With Chronic Traumatic Brain Injury Symptoms Throughout a Full-time or Part-time Holistic Cognitive Rehabilitation Program: An Initial Assessment.
Brief Title: Assessing Brain Changes Throughout the ABI Wellness Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: NeuroCatch Platform became commercially available (Health Canada License approved) and can now be incorporated into the ABI Wellness Program
Sponsor: NeuroCatch Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NCI_CogRehab_001
Record Dates: First submitted 2018-01-23; First posted 2018-02-20 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Brain Injuries
MeSH Terms: conditions — Brain Injuries

STUDY DESIGN:
Intervention Model Description: Participants will self-select into one of two treatment conditions: a full-time intensive program or a part-time program. Participants in the full-time program will be asked to complete 4 experimental sessions with the NeuroCatch PlatformTM over the course of 3 months (i.e. one session/ month); whereas, participants in the part-time program will be asked to complete 3 scans over 3 months (i.e. one session/1.5 months).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full-time Cognitive Rehabilitation Program (Experimental): Participants in full-time program will be asked to complete 4 experimental sessions with the NeuroCatch Platform™ over the course of 3 months (i.e. one session/ month).
  Interventions: Device: NeuroCatch Platform™
- Part-time Cognitive Rehabilitation Program (Experimental): Participants in the part-time program will be asked to complete 3 experimental sessions with the NeuroCatch Platform™ over 3 months (i.e. one session/1.5 months).
  Interventions: Device: NeuroCatch Platform™

INTERVENTIONS:
Device: NeuroCatch Platform™ — NeuroCatch Platform™ consists of software and hardware that captures brain health information. The platform intends to provide a quick, portable and easy to use solution for the acquisition, display, analysis, storage, reporting and management of electroencephalograph (EEG) and event-related potential (ERP) information.

SUMMARY:
Symptoms resulting from mild/moderate trauma to the brain are as varied as the individuals who sustain them. The currently held belief is that the majority of healing and functional recovery occurs within the first two years post injury. A large proportion of individuals who sustain mild/moderate brain injuries (mTBIs) do not fully recover, and continue to experience symptoms well beyond two years post injury. Cognitive rehabilitation programs have been shown to be somewhat effective in helping mTBI patients regain some functionality in these executive domains.

The purpose of the current study is to use an objective assessment of brain function to track changes during either a full-time or part-time holistic cognitive rehabilitation program, specifically the ABI Wellness (ABIW) program. The NeuroCatch Platform™ test will be used to assess brain functioning before, during and after 3 months in the ABIW program. The NeuroCatch Platform™ test uses electroencephalography (EEG) to measure event-related potential (ERP) signals produced by the brain, in response to an auditory stimulus. Three brain processes are examined with this test: Auditory sensation (ERP marker is the N100), Basic attention (ERP marker is the P300), and Cognitive processing (ERP marker is the N400).

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in but not initiated the ABI Wellness program
2. Male or female, 19-65 years old inclusively
3. Normal hearing capabilities
4. Able to understand the informed consent form, study procedures and willing to participate in study
5. Able to keep eyes still for 6 minutes

Exclusion Criteria:

1. Clinically documented hearing issues (e.g. in-ear hearing problems, punctured ear drum, etc.)
2. Score of 7 or lower on the Mini Mental State Exam (MMSE) - Orientation subscale
3. Implanted pacemaker
4. Metal or plastic implants in skull
5. In-ear hearing aid or cochlear implant, hearing device
6. Recent (within last 6 months) acquired brain injury
7. History of other neurological disorder (e.g. brain cancer, dementia, multiple sclerosis, stroke, etc.)
8. Exposed to investigational drug or device 30 days prior to start in this study, or concurrent use of investigational drug or device while enrolled in this study
9. Not fluent in English language
10. Unable to provide informed consent
11. Previous participation in studies using the NeuroCatch Platform™
12. If female and of child-bearing potential: pregnant, suspected or planning to become pregnant or breast-feeding
13. History of seizures
14. Allergy to rubbing alcohol or EEG gel

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2020-04-21 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Tracking and comparison of neurophysiological changes (response size) to functional changes as participants complete 3 months of the ABIW program. | 3 months
  Response size will be measured as amplitude in microvolts. Functional changes will be measured using a proprietary BrainEx Assessment that provides a category score from four cognitive programs of BrainEx.
Tracking and comparison of neurophysiological changes (response timing) to functional changes as participants complete 3 months of the ABIW program. | 3 months
  Response timing will be measured as latency in milliseconds. Functional changes will be measured using a proprietary BrainEx Assessment that provides a category score from four cognitive programs of BrainEx.

SECONDARY OUTCOMES:
Collection and evaluation of adverse events and adverse device effects | 3 months
  Evaluate the tolerability and performance of the NeuroCatch Platform™ with individuals who have chronic cognitive deficits due to traumatic brain injury.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Venter, MBChB MFamMed CCFP IFMCP, Principal Investigator — HealthTech Connex Inc. Centre for Neurology Studies
Locations (1):
- HealthTech Connex Inc. Centre for Neurology Studies, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided